CLINICAL TRIAL: NCT00957385
Title: A Randomized Phase II Study of Lenalidomide Maintenance Therapy in AML Patients Aged > 60 Years in CR1 or Higher and < 60 Years in CR2 or Higher
Brief Title: Maintenance Therapy in Acute Myeloid Leukemia (AML) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV-AML-PI-166
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2009-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Leukemia; Remission
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Arm A will receive Revlimid.
  Interventions: Drug: Revlimid
- B (No Intervention): Arm B will not receive Revlimid but an observational arm

INTERVENTIONS:
Drug: Revlimid — 10mgs PO daily for 21 days of each 28 day cycle. Number of cycles: total of 24 or until subject relapses or unacceptable toxicity develops.
  Other Names: Lenalidomide
  Arms: A

SUMMARY:
The purpose of this study is to determine if Revlimid will help maintain patients with acute myeloid leukemia in remission.

DETAILED DESCRIPTION:
At present, the majority of AML patients >60 years of age that achieve CR and thereafter successfully complete further chemotherapy, are not candidates for allogeneic bone marrow transplantation (alloBMT) due to their age. Rather, this group of patients is simply observed until relapse occurs. In this age group, the median duration of CR is only ~10 months. The survival of patients <60 years of age who are not candidates for transplantation (due to donor unavailability), and who are in CR2 or higher is also extremely poor. Several lines of evidence suggest that the immune system - and in particular AML specific CTLs and NK cells - is capable of recognizing and clearing AML cells.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute myeloid leukemia in remission.
* Able to take aspirin 81mgs daily.

Exclusion Criteria:

* Pregnant or breast feeding females.
* Known hypersensitivity to thalidomide.
* Any prior use of lenalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility and assess the effect on relapse free survival by giving Revlimid in the post complete remission maintenance setting | The 1st interim analysis will be done once all subjects have completed 12 cycles, and the 2nd interim analysis will be done once all subjects have completed treatment.

SECONDARY OUTCOMES:
To determine the toxicity of Revlimid when given in the maintenance setting. | The 1st interim analysis will be done after all subjects have receieved 12 cycles and the 2nd when all subjects have completed treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Andre Schuh, MD.FRCP(C), Principal Investigator — University Health Network Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada